CLINICAL TRIAL: NCT03587610
Title: Evaluation of a Tdap-IPV Vaccination Remedial Strategy on Vaccination Coverage in Patients 65 Years of Age or Older in the French County of Sarthe
Brief Title: Evaluation of a Tdap-IPV (Tetanus, Diphteria, Pertussis and Inactivated Polio) Vaccination Remedial Strategy on Vaccination Coverage in Patients 65 Years of Age or Older
Acronym: HOSPIVAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHM-2017-S6/06
Record Dates: First submitted 2018-06-21; First posted 2018-07-16 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2018-07

CONDITIONS: Vaccination
Keywords: vaccination coverage

STUDY DESIGN:
Intervention Model Description: Single center, prospective, cluster randomized trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): * if the patients vaccinations are up to date: no remedial vaccination is done and the patient is informed of the next remedial vaccination date
  * if the patients vaccinations are not up to date: remedial vaccination is realised in the unit in the absence of contraindication, in case of a temporary contraindication the vaccination will be performed on an outpatient basis by the patients primary care provider and he will be given a prescription at hospital discharge for the remedial vaccination.
  Interventions: Biological: Remedial vaccination
- Standard care (No Intervention): * if the patients vaccinations are up to date: no remedial vaccination is done and the patient is informed of the next remedial vaccination date
  * if the patients vaccinations are not up to date: the patient will be informed that a remedial vaccination is necessary and that he should contact his primary care provider after hospital discharge.

INTERVENTIONS:
Biological: Remedial vaccination — * if the patients vaccinations are up to date: no remedial vaccination is done and the patient is informed of the next remedial vaccination date
  * if the patients vaccinations are not up to date: remedial vaccination is realised in the unit in the absence of contraindication, in case of a temporary contraindication the vaccination will be performed on an outpatient basis by the patients primary care provider and he will be given a prescription at hospital discharge for the remedial vaccination.
  Arms: Intervention arm

SUMMARY:
In France, vaccination coverage is insufficient (in 2002, 71.2% coverage for tetanus, 41.9% for poliomyelitis and 33.7% for diphteria). These numbers decrease significantly with age: coverage for people aged over 65 was 60.5%, 13.3% and 10.5% for tetanus, poliomyelitis and diphteria coverage respectively.

The primary objective of this study is to evaluate the impact of a hospital based vaccination remedial strategy for Tdap-IPV (tetanus, diphteria, pertussis and polio vaccine) in patients 65 years of age or older.

Secondary objectives are to measure the vaccination coverage of patients aged 65 years or older hospitalised in a medical ward in our hospital, to evaluate their knowledge of their vaccination coverage, and to evaluate the socio-demographic factors associated with vaccination coverage.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years or older
* Patients capable of understanding and giving informed consent to participate in the study
* Valid social security coverage

Exclusion Criteria:

* Patients under judicial safeguard measures
* Refusal to participate in the study
* Vaccination contra-indication
* Patient already included in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2018-05-24 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change in immunization rate after a hospital centered remedial strategy for Tdap-IPV vaccination in patients 65 years or older | two months
  Difference in the increase in vaccination coverage between the two arms, measured as a percentage

SECONDARY OUTCOMES:
Immunisation rate among patients 65 years of age or older in the Sarthe department of France | two months
  Pre-intervention vaccination coverage rate in both arms, measured as a percentage
Immunisation rate according to sex among patients 65 years or older | two months
  Sex of patients included in the study
Immunisation rate according to primary care coverage among patients 65 years of age or older | two months
  Primary care coverage is defined as having a regular primary care physician registered as such with French social security.
Immunisation rate according to socio professional category | two months
  Socio professional category defined according to the French national institute for statistics and economic studies (INSEE)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Blanchi, M.D., Principal Investigator — Centre Hospitalier du Mans
Locations (1):
- Centre Hospitalier Le Mans, Le Mans, France

IPD SHARING:
Plan to Share IPD: Undecided